CLINICAL TRIAL: NCT02526953
Title: Randomised Phase III Trial of Chemoradiotherapy With or Without Paclitaxel in Patients With Squamous-cell Anal Cancer
Brief Title: Efficacy Study of Chemoradiotherapy With or Without Paclitaxel in Squamous-cell Anal Carcinoma Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Blokhin's Russian Cancer Research Center (Other)
Responsible Party: Principal Investigator, Sergey Gordeyev, Principal Investigator, Blokhin's Russian Cancer Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCAC-001
Record Dates: First submitted 2015-08-15; First posted 2015-08-18 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Anus Neoplasms; Carcinoma, Squamous Cell; Anus Diseases; Neoplasms; Neoplasms, Squamous Cell; Carcinoma
Keywords: anal cancer; chemoradiation; intensity-modulated radiotherapy; paclitaxel
MeSH Terms: conditions — Anus Neoplasms; Carcinoma, Squamous Cell; Anus Diseases; Neoplasms; Neoplasms, Squamous Cell; Carcinoma | interventions — Paclitaxel; Capecitabine; Mitomycins; Mitomycin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paclitaxel (Experimental): Patients will receive intensity-modulated radiotherapy with dose based on T stage. The planned doses to the primary tumor and pelvis are 52-58 Gy and 44 Gy, respectively.The concurrent chemotherapy regimen will consist of paclitaxel 45 mg/m2 on days 3,10,17,24,31, capecitabine 625 mg/m2 bid on treatment days and mitomycin C 10 g/m2 on day 1.
  Interventions: Drug: Paclitaxel; Drug: Capecitabine; Drug: Mitomycins; Radiation: Radiotherapy
- Standard (Active Comparator): Patients will receive intensity-modulated radiotherapy with dose based on T stage. The planned doses to the primary tumor and pelvis are 52-58 Gy and 44 Gy, respectively.The concurrent chemotherapy regimen will consist of capecitabine 825 mg/m2 bid on treatment days and mitomycin C 12 g/m2 on day 1.
  Interventions: Drug: Capecitabine; Drug: Mitomycins; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel — 45 mg/m2, IV, weekly during the radiation. Number of infusions: 5.
  Other Names: (2α,4α,5β,7β,10β,13α)-4,10-bis(acetyloxy)-13-{[(2R,3S)- 3-(benzoylamino)-2-hydroxy-3-phenylpropanoyl]oxy}- 1,7-dihydroxy-9-oxo-5,20-epoxytax-11-en-2-yl benzoate
  Arms: Paclitaxel
Drug: Capecitabine — 625 mg/m2, bid, per os, only on days of radiation (Monday through Friday)
  Other Names: Xeloda
  Arms: Paclitaxel
Drug: Capecitabine — 825 mg/m2, bid, per os, only on days of radiation (Monday through Friday)
  Other Names: Xeloda
  Arms: Standard
Drug: Mitomycins — 10 mg/m2, IV, on day 1. Number of infusions: 1.
  Other Names: Mitomycin C; MMC
  Arms: Paclitaxel
Drug: Mitomycins — 12 mg/m2, IV, on day 1. Number of infusions: 1.
  Other Names: Mitomycin C; MMC
  Arms: Standard
Radiation: Radiotherapy — Dose: 44 Gy on regional nodes, 52-58 Gy on primary tumor, based on T stage

SUMMARY:
The purpose of this study is to determine whether the combination of paclitaxel, capecitabine, mitomycin and intensity-modulated radiotherapy is more effective than the standard combination of capecitabine, mitomycin and intensity-modulated radiotherapy (IMRT) in patients with squamous-cell anal cancer.

DETAILED DESCRIPTION:
This trial aims to investigate the efficacy of chemoradiotherapy with or without paclitaxel in squamous-cell anal cancer. This is a prospective multicenter open-label randomized phase III clinical trial. Patients will be randomized using an online randomization system to receive either standard IMRT with capecitabine and mitomycin or IMRT with capecitabine, mitomycin and paclitaxel. A stratification will be performed based on T stage, N stage and clinical center. Doses of capecitabine and mitomycin in experimental group were reduced for better treatment tolerance. The target accrual is 157 patients in each treatment arm (including 10% potential data loss) based on potential benefit of 15% 3-yr disease-free survival (70% vs 85%), α=0,05, power 80% in the experimental arm. An interim analysis is planned after 50% of the patients will reach a 3-year followup. Pelvic Magnetic Resonance Imaging (MRI) is performed in all patients for staging and followup. Pelvic MRI and histological diagnosis are subject to central review. Conduction of this study and data collection are controlled by a local institutional board.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Histologically verified squamous-cell anal cancer
* Stage I-IIIB (Union for International Cancer Control (UICC) TNM classification v7)
* Eastern Cooperative Oncology Group (ECOG) status 0-2
* HIV (Human Immunodeficiency Virus) negative
* Haemoglobin (HGB) > 90 g/L
* Platelet Count (PLT) > 120x10*9/L
* Serum creatinine < 150 µmol/L
* Total bilirubin < 25 µmol/L

Exclusion Criteria:

* inability to obtain informed consent
* distant metastases
* synchronous or metachronous tumors
* previous chemotherapy or radiotherapy
* clinically significant cardiovascular disorders (myocardial infarction < 6 months before visit, stroke < < 6 months before visit, instable angina < 3 months before visit, arrhythmia, uncontrolled hypertension > 160/100 mm hg
* clinically significant neurological disorders
* previous neuropathy 2 or higher
* current infection or heavy systemic disease
* pregnancy, breastfeeding
* ulcerative colitis
* individual intolerance to treatment components
* proven dihydropyrimidine dehydrogenase (DPD) deficiency
* participation in other clinical trials
* psychiatric disorders, which render patient unable to follow instructions or understand his/her condition
* technical inability to perform pelvic MRI
* inability of long-term followup of the patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years

SECONDARY OUTCOMES:
Complete response at 26 weeks | 26 weeks
3-year colostomy-free survival | 3 years
3-year cancer-specific survival | 3 years
3-year overall survival | 3 years
Acute toxicity measured according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v.4.0 | 30 days
  Toxicity measured according to NCI-CTCAE v.4.0
Late toxicity measured according to Radiation Therapy Oncology Group (RTOG) criteria | 3 years
  Late toxicity measured according to RTOG criteria

OTHER OUTCOMES:
Quality of life according to European organization for research and treatment of cancer (EORTC) Quality of Life questionnaire (QLQ)-C30 (v.3) scale | 3 years
  Change from baseline in quality of life on the EORTC QLQ-C30 (v.3) scale

CONTACTS AND LOCATIONS:
Overall Officials: Arsen O Rasulov, PhD, Study Chair — N.N.Blokhin Russian Cancer Research Center